CLINICAL TRIAL: NCT05215002
Title: Quality Assurance Via Telephone Interviews After Cataract Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Cat Tel
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Cataract
Keywords: Telephone Call
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telephone call (Experimental): Patient will receive a telephone call in the evening of the day of the surgery or one day after surgery
  Interventions: Other: Telephone Call
- No telephone call (Experimental): Patient will not receive a telephone call in the evening of the day of the surgery or one day after surgery
  Interventions: Other: No telephone call

INTERVENTIONS:
Other: Telephone Call — Patient will be called in the evening of the day of the surgery or one day after surgery and asked about any complaints
  Arms: Telephone call
Other: No telephone call — Patient will not be called in the evening of the day of the surgery or one day after surgery and asked about any complaints
  Arms: No telephone call

SUMMARY:
To analyse quality assurance after cataract surgery by assessing discomfort and other symptoms via telephone interviews either in the evening of the day of the surgery or 1 day after surgery versus no additional call after surgery.

DETAILED DESCRIPTION:
As there is a trend towards shorter hospital stays, an increasing number of patients is leaving the hospital the same day after cataract surgery. There may be questions or complaints after the patients' dismissal after cataract surgery, consequently it might be useful to call patients at the day or one day after surgery in order to ask them about their concerns.

In general, possible complications after cataract surgery are explained to patients already before surgery and patients often receive additional written information. But as patients may still be uncertain whether it would be beneficial to visit a doctor in case of problems, it might be useful to call the patients and if necessary, advise them to see a doctor. During the phone call patients have the opportunity to ask more questions if something still does not seem clear.

For patients who are scheduled for cataract surgery for both eyes, the routine procedure is as follows: if cataract surgery is scheduled for both eyes, in general the surgeries are performed one week apart. Cataract surgery is usually performed under local anaesthesia and the patient can leave the department on the same day. When patients arrive at the department of ophthalmology for the second surgery, doctors evaluate the condition of the eye, operated the week before. After each surgery of each eye patients receive a prescription of topical medication. It is recommended to see the referring ophthalmologist within a week after the procedure. In case of problems or complaints patients are always told to see a doctor immediately. A respective written information is given to the patients.

During this study we plan to call patients, who are scheduled for cataract surgery for both eyes, in the evening of the day of the surgery or one day after the surgery of the first eye and to ask questions about their current condition for quality assessment. When people return for cataract surgery of the second eye, a questionnaire will be handed out to the patients. This questionnaire includes questions concerning problems after surgery of the first eye, visits in outpatint clinics and about their satisfaction with the phone call after the surgery of the first eye.

In this study 200 patients will be included: 100 patients will receive a telephone call (50 in the evening of the day of the surgery, 50 one day after surgery) and 100 patients who will not receive a phone call.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged 18 and older
* planned cataract surgery of both eyes
* good knowledge of the german language

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-11-19 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients | 24 months
  The number of patients in group 1 and group 2 seen at the outpatient clinic between surgery of the first and the second eye will be documented

SECONDARY OUTCOMES:
Patient's Satisfaction | 24 months
  Patient's satisfaction with the telephone call after cataract surgery will be assessed with a question asking the patient if she/ he liked the call (5 answering options: very, a little, I don't know, no, absolutely not)
Patient's Symptoms | 24 months
  Patient's symptoms after cataract surgery will be assessed during the telephone interview and the questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, MD, Principal Investigator — Vienna Institute for Research in Ocular Surgery
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Hanusch Hospital, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No